CLINICAL TRIAL: NCT04743297
Title: Labour Induction With the Propess Vaginal Delivery System vs. Labour Induction With the Prostin Vaginal Tablet in Case of a Prelabour Rupture of Membranes. PESTIBOR Randomized Controlled Trial
Brief Title: Propess Versus Prostin for Induction of Labour in Women With Term PROM
Acronym: PESTIBOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRP-2020/01-04
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Premature Rupture of Membranes at Term; Induction of Labour
Keywords: Induction; PROM; Propess; Prostin
MeSH Terms: interventions — Dinoprostone; KLK15 protein, human

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propess Vaginal Delivery System (Active Comparator): Propess - Prostaglandin E2 Vaginal Delivery System. Slow intravaginal release of 10 mg dinoprostone at a rate of 0.3 mg/h.
  Interventions: Drug: Prostaglandin E2 (Propess)
- Prostin Tablet (Active Comparator): Prostaglandin E2 Vaginal Tablet 3 mg dinoprostone
  Interventions: Drug: Prostaglandin E2 (Prostin)

INTERVENTIONS:
Drug: Prostaglandin E2 (Propess) — Propess - The vaginal insert is removed 24 h after the application. It is only to be removed earlier in case of the onset of active labour or at the occurrence of hyperstimulation.
  Other Names: dinoprostone
  Arms: Propess Vaginal Delivery System
Drug: Prostaglandin E2 (Prostin) — Prostin - 3 mg vaginal tablet is placed in the posterior vaginal fornix. Dose can be repeated every 8 hours till onset of active labour or the occurrence of hyper-stimulation.
  Other Names: dinoprostone
  Arms: Prostin Tablet

SUMMARY:
Premature rupture of membranes (PROM) at term is a rupture that occurs at term (> 37 weeks) before the start of labor.

The purpose of the study was to compare the safety and efficacy of two agents used in induction of labor in women with term PROM Propess (Controlled release dinoprostone, Vaginal Delivery System) and Prostin E2 (Dinoprostone vaginal Tablet).

Women will be randomised to two treatment groups.

Although some studies support efficacy of the Propess for cervical ripening at term in induction of labor with intact membranes, it has not been well studied in women with PROM at term.

DETAILED DESCRIPTION:
The study is going to include all pregnant women with in-term PROM (after week 37 of pregnancy) without contractions if they meet the inclusion criteria. If the cervix is still non-inducible after 4-6 hours and there are no contractions, the medication to be administered to them will be determined by means of computer randomization. The success rate of induction with Propess vs. Prostin tablets will be compared. Soon after PROM, there can be the onset of contractions and cervix dilation that lead to childbirth.

In case of some pregnant women, there are no contractions and cervix dilation even after the event despite PROM and water breaking. If the status remains unchanged, the risk of intrauterine infection, fetus infection, and later on an infection of the newborn increases. The expecting mother can also eventually lose hope for a successful vaginal birth and starts thinking about having a caesarean delivery. To avoid that, the investigators use medications that accelerate the onset of vaginal birth in clinical practice.

The investigators know several ways to induce labour after PROM. References give no clear and reliable data on the best approach. The investigators can use medications such as oxytocin, dinoprostone, or misoprostol.

Our ward has been using Prostin 3 mg (dinoprostone) vaginal tablets to induce labour in case of PROM for several years. They have proven to be an efficient and safe procedure in our clinical practice.

Propess is used for the induction of labor with intact membranes. Based on the information from references and according to our experience, the medication is highly effective and safe, as well as easy to use.

Our study aims at establishing whether it can also be used with pregnant women with PROM.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Gestational age 37 weeks or more
* Singleton pregnancy
* Cephalic presentation
* Unfavorable cervix (BISHOP <6)
* No contraindications for vaginal delivery
* Without uterine surgery
* Without chorioamnionitis

Exclusion Criteria:

* Age less than 18 years
* Multiple gestation
* Previous cesarean section
* Suspected intraamniotic infection
* Any contraindication to vaginal delivery
* Bishop score >7
* Pathological ctg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 526 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Induction to Delivery Interval | 24 hours
Induction to Onset of labor Interval | 24 hours

SECONDARY OUTCOMES:
Frequency of Cesarean Sections | 24 hours
Frequency of Failed Induction | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Anzeljc, Study Chair — Maribor University Medical Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mynarek M, Bjellmo S, Lydersen S, Strand KM, Afset JE, Andersen GL, Vik T. Prelabor rupture of membranes and the association with cerebral palsy in term born children: a national registry-based cohort study. BMC Pregnancy Childbirth. 2020 Jan 31;20(1):67. doi: 10.1186/s12884-020-2751-3. PMID 32005186
- [Background] National Collaborating Centre for Women's and Children's Health. National Institute for Health and Care Excellence: Clinical Guidelines. Intrapartum Care: Care of Healthy Women and Their Babies During Childbirth. London: National Institute for Health and Care Excellence (UK) Copyright (c) 2014 National Collaborating Centre for Women's and Children's Health.; 2014
- [Background] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Background] Zlatnik FJ. Management of premature rupture of membranes at term. Obstet Gynecol Clin North Am. 1992 Jun;19(2):353-64. PMID 1630743
- [Background] Geethanath RM, Ahmed I, Abu-Harb M, Onwuneme C, McGarry K, Hinshaw K. Intrapartum antibiotics for prolonged rupture of membranes at term to prevent Group B Streptococcal sepsis. J Obstet Gynaecol. 2019 Jul;39(5):619-622. doi: 10.1080/01443615.2018.1550474. Epub 2019 Mar 27. PMID 30917724
- [Background] Ivars J, Garabedian C, Devos P, Therby D, Carlier S, Deruelle P, Subtil D. Simplified Bishop score including parity predicts successful induction of labor. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:309-14. doi: 10.1016/j.ejogrb.2016.06.007. Epub 2016 Jul 5. PMID 27423032
- [Background] Athiel Y, Crequit S, Bongiorno M, Sanyan S, Renevier B. Term prelabor rupture of membranes: Foley catheter versus dinoprostone as ripening agent. J Gynecol Obstet Hum Reprod. 2020 Oct;49(8):101834. doi: 10.1016/j.jogoh.2020.101834. Epub 2020 Jun 22. PMID 32585393
- [Background] Freret TS, Chacon KM, Bryant AS, Kaimal AJ, Clapp MA. Oxytocin Compared to Buccal Misoprostol for Induction of Labor after Term Prelabor Rupture of Membranes. Am J Perinatol. 2021 Feb;38(3):224-230. doi: 10.1055/s-0039-1696642. Epub 2019 Sep 6. PMID 31491801
- [Background] Cheung PC, Yeo EL, Wong KS, Tang LC. Oral misoprostol for induction of labor in prelabor rupture of membranes (PROM) at term: a randomized control trial. Acta Obstet Gynecol Scand. 2006;85(9):1128-33. doi: 10.1080/00016340600589636. PMID 16929421
- [Background] Hu YP, Zhou D, Li M, Wang Y, Wang L, Sun GQ, Xiao M. Use of labor induction with dinoprostone vaginal suppositories in pregnant women with gestational hypertension. J Obstet Gynaecol Res. 2019 Nov;45(11):2185-2192. doi: 10.1111/jog.14092. Epub 2019 Aug 27. PMID 31456315
- [Background] Shirley M. Dinoprostone Vaginal Insert: A Review in Cervical Ripening. Drugs. 2018 Oct;78(15):1615-1624. doi: 10.1007/s40265-018-0995-2. PMID 30317521
- [Background] Pajntar M, Lučovnik M. Normalni porod in vodenje poroda. v knjigi Nosečnost in vodenje poroda. Ured. Pajntar M, Novak Antolič Ž, Lučovnik M. Medicinski razgledi 2015. Tretja dopolnjena izdaja. 231-50.